CLINICAL TRIAL: NCT04969679
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Effect of Mutaflor in Patients With Mild-to-moderate Ulcerative Colitis on 5-ASA Treatment.
Brief Title: Additive Effect of Probiotics (Mutaflor®) in Patients With Ulcerative Colitis on 5-ASA Treatment.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Soo-kyung Park, Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MUTAUC01
Record Dates: First submitted 2021-07-07; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Ulcerative Colitis
Keywords: Mutaflor
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E. coli Nissle 1917 (Mutaflor®) (Active Comparator): Active group will receive E. coli Nissle 1917 (Mutaflor®).
  Interventions: Drug: E. coli Nissle 1917 (Mutaflor®)
- Placebo (Placebo Comparator): Placebo group will receive placebo drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E. coli Nissle 1917 (Mutaflor®) — Take 1 capsule per day in the morning from the first day to the fourth day and take 2 capsules per day from the fifth day to the end of the testing period.(for 8 weeks)
  Arms: E. coli Nissle 1917 (Mutaflor®)
Drug: Placebo — Take 1 capsule per day in the morning from the first day to the fourth day and take 2 capsules per day from the fifth day to the end of the testing period.(for 8 weeks)
  Arms: Placebo

SUMMARY:
E.coli Nissle 1917 (Mutaflor®) is equivalent to mesalazine in preventing disease relapse in ulcerative colitis. However, data on ability of E.coli Nissle 1917 (Mutaflor®) to induce remission compared with placebo is limited. Investigators aim to investigate the efficacy of E.coli Nissle 1917 (Mutaflor®) as an add-on treatment to 5-ASA in mild to moderate ulcerative colitis.

DETAILED DESCRIPTION:
This is a multicentre, double-blind, randomised, placebo-controlled study in patients with mild-to-moderate UC.

Subjects were randomly assigned to receive either E.coli Nissle 1917 (Mutaflor®) or placebo once daily for 8 weeks, and inflammatory bowel disease questionnaire (IBDQ) scores, clinical remission, and response rate were compared.

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative colitis patients over the age of 19 with mild to moderate symptoms using 5-ASA (Mayo score 3-9)
* Patient who signed the consent form

Exclusion Criteria:

* The extent of ulcerative colitis is limited to proctitis
* History of bowel resection
* History of using other medication than 5-ASA such as immunomodulators, steroid or biologics within 3months
* history of using antibiotics or probiotics within 2 weeks
* Pregnant or lactating woman
* Requiring hospitalization and imminent need for surgery

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2020-06-03 (Actual)

PRIMARY OUTCOMES:
Compare and evaluate the increase in IBDQ(Inflammatory bowel disease questionnaire) score between the Mutaflor group and the Placebo group | 8weeks
  The evaluation of the beneficial effects of Mutaflor on mild-to-moderate UC patients, was assessed by an increase in the IBDQ score more than 16 points from baseline to week 8.
  The Score can range from 32 to 224, with higher scores reflecting better HRQOL(Health-related quality of life)

SECONDARY OUTCOMES:
Evaluate the clinical remission between Mutaflor group and Placebo group | 4weeks, 8weeks
  Partial Mayo≤1, assessed at week 4 or Mayo≤2, assessed at week 8. Mayo score can range from 0-12 with higher scores indicating worse severity.
Evaluate the clinical response between Mutaflor group and Placebo group | 4weeks, 8weeks
  Partial Mayo≤2 or decrease more than 2 points, assessed at week 4 or Mayo≤ 2 or decrease more than 2 points, assessed at week 8.
  Mayo score can range from 0-12 with higher scores indicating worse severity.
Improvement in endoscopic scores between Mutaflor group and Placebo group | 8weeks
  Assessed by the endoscopic subgroup score=0 of the mayo. Mayo Endoscopic Sub Scores can range from 0-3, with higher scores indicating worse severity.
Evaluate the endoscopic response between Mutaflor group and Placebo group | 8weeks
  Assessed by the endoscopic subgroup score=0 or decrease more than 1 point. Mayo Endoscopic Sub Scores can range from 0-3 with higher scores indicating worse severity.
Evaluate the Microbiome(stool) change between Mutaflor group and Placebo group | 8weeks
  Stool microbial change including diversity. DNA extraction from stool samples and 16S rRNA gene sequencing analysis. calculating α- and β-diversities.

CONTACTS AND LOCATIONS:
Locations (1):
- Soo-kyung Park, Seoul, South Korea

REFERENCES:
- [Derived] Park SK, Kang SB, Kim S, Kim TO, Cha JM, Im JP, Choi CH, Kim ES, Seo GS, Eun CS, Han DS, Park DI. Additive effect of probiotics (Mutaflor) on 5-aminosalicylic acid therapy in patients with ulcerative colitis. Korean J Intern Med. 2022 Sep;37(5):949-957. doi: 10.3904/kjim.2021.458. Epub 2022 Mar 31. PMID 36068716